CLINICAL TRIAL: NCT06575543
Title: Anatomical Transportal ACL Reconstruction : Effect of Using 2 or 3 Portal Technique on Femoral Tunnel Position
Brief Title: CT Evaluation of ACL Anatomical Reconstruction
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Almeldien Mohamed, Dr, Assiut University
Other Study IDs: CT evaluation of ACL repair
Record Dates: First submitted 2024-08-24; First posted 2024-08-28 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2 portal group: The conventional 2-portal technique uses the anterolateral portal as the viewing portal and the anteromedial portal as the working portal
  Interventions: Radiation: CT
- 3 portal group: the 3-portal technique allows interchangeable use of the portals as a viewing and working portals depending on the specific task that is being performed
  Interventions: Radiation: CT

INTERVENTIONS:
Radiation: CT — 3D CT scan have been used to evaluate the tunnels location after ACL reconstruction, as they can provide excellent perspective of the tunnel aperture, good visualization of bony structure and shape of the intercondylar notch, that preclude the use of a conventional 2-dimensional CT scan for measurement of the ACL tunnels location

SUMMARY:
Our research is to evaluate the position and length of femoral tunnel, and to examine whether knee stability and clinical functional outcomes are better while using two-portal or three-portal technique .

DETAILED DESCRIPTION:
Arthroscopic anterior cruciate ligament (ACL) reconstruction is one of the most often performed orthopedic surgeries . Restoration of normal anatomy after ACL reconstruction is related to achieve better function and a satisfactory long-term outcomes. The principles for anatomical ACL reconstruction are to functionally reestablish the ACL to its native dimensions, collagen orientation and insertion sites . The basis for the completion of these principles lies in the correct identification of the insertion sites. The conventional 2-portal technique uses the anterolateral portal as the viewing portal and the anteromedial portal as the working portal. the 3-portal technique allows interchangeable use of the portals as a viewing and working portals depending on the specific task that is being performed. The internal joint anatomy, as soft tissue remnants and bony landmarks, should guide the placement of the portals in ACL anatomical reconstruction and that each of the portals has a specific role during ACL anatomical reconstruction . So does the improved visualization through 3-portal technique compared to 2-portal technique have an impact on femoral tunnel position ?

ELIGIBILITY:
Inclusion Criteria:

1. Age ( 16 - 50 ) .
2. Isolated ACL tear with or without meniscal inj
3. Patient who have undergone ACL reconstruction in the last 5 years in Arthroscopy and sports injuries unit .

Exclusion Criteria:

* 1- Age ( < 16 ) 2- Patient with multi ligamentous inj . 3- Revision ACL tear .

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Postoperative evaluation of patients who had previous ACL reconstruction (within terms of inclusion criteria & study sample ) by ct , clinical examination and functional scores .
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Ct evaluation | 1 day after surgery
  3D CT scan have been used to evaluate the tunnels location after ACL reconstruction, as they can provide excellent perspective of the tunnel aperture, good visualization of bony structure and shape of the intercondylar notch, that preclude the use of a conventional 2-dimensional CT scan for measurement of the ACL tunnels location

SECONDARY OUTCOMES:
Clinical Examination & Functional scores | at least 2 years after surgery
  - KOOS ( Knee Injury & Osteoarthritis Outcome ) The KOOS's five patient-relevant dimensions are scored separately: Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No problems) to 4 (Extreme problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Lohmander LS, Ostenberg A, Englund M, Roos H. High prevalence of knee osteoarthritis, pain, and functional limitations in female soccer players twelve years after anterior cruciate ligament injury. Arthritis Rheum. 2004 Oct;50(10):3145-52. doi: 10.1002/art.20589. PMID 15476248
- [Background] Bedi A, Altchek DW. The "footprint" anterior cruciate ligament technique: an anatomic approach to anterior cruciate ligament reconstruction. Arthroscopy. 2009 Oct;25(10):1128-38. doi: 10.1016/j.arthro.2009.03.008. Epub 2009 Aug 22. PMID 19801292
- [Background] van Eck CF, Schreiber VM, Liu TT, Fu FH. The anatomic approach to primary, revision and augmentation anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2010 Sep;18(9):1154-63. doi: 10.1007/s00167-010-1191-4. Epub 2010 Jun 9. PMID 20532865
- [Background] Nikolaou VS, Efstathopoulos N, Sourlas I, Pilichou A, Papachristou G. Anatomic double-bundle versus single-bundle ACL reconstruction: a comparative biomechanical study in rabbits. Knee Surg Sports Traumatol Arthrosc. 2009 Aug;17(8):895-906. doi: 10.1007/s00167-009-0754-8. Epub 2009 Mar 17. PMID 19290508
- [Background] Snow M, Stanish WD. Double-bundle ACL reconstruction: how big is the learning curve? Knee Surg Sports Traumatol Arthrosc. 2010 Sep;18(9):1195-200. doi: 10.1007/s00167-010-1062-z. Epub 2010 Feb 6. PMID 20140602